CLINICAL TRIAL: NCT02350634
Title: A High Resolution Autopsy Study Evaluating the Relationship of 18F-AV-1451 PET Imaging and Tau Pathology
Brief Title: 18F-AV-1451 High Resolution Autopsy Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A13
Record Dates: First submitted 2015-01-08; First posted 2015-01-30 (Estimated); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autopsy Cohort (Experimental): End-of-life subjects (life expectancy < 6 months) consenting to brain donation at autopsy. Subjects will receive a single IV bolus injection of 370 MBq(10 mCi) of flortaucipir F18.
  Interventions: Drug: Flortaucipir F18

INTERVENTIONS:
Drug: Flortaucipir F18 — Subjects will receive a single IV bolus injection of 370 megabecquerel (MBq) (10 millicurie [mCi]) of flortaucipir.
  Other Names: [F-18]T807; 18F-AV-1451

SUMMARY:
The study is designed to examine the relationship between imaging results detected on a 18F-AV-1451 PET scan and pathology found at autopsy within six months of imaging.

ELIGIBILITY:
Inclusion Criteria:

* Projected life expectancy ≤ 6 months

Exclusion Criteria:

* Primary brain tumor, known metastases to the brain, central nervous system lymphoma
* Major, focal structural brain lesion
* Aggressively being treated with life sustaining measures
* Clinically significant infectious disease
* History of risk factors for Torsades de Pointes or are currently taking medication known to cause QT prolongation
* Have received or participated in a trial with investigational medications in the past 30 days
* Females of childbearing potential who are pregnant or not using adequate contraception

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-11-26 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Ushizima D, Chen Y, Alegro M, Ovando D, Eser R, Lee W, Poon K, Shankar A, Kantamneni N, Satrawada S, Junior EA, Heinsen H, Tosun D, Grinberg LT. Deep learning for Alzheimer's disease: Mapping large-scale histological tau protein for neuroimaging biomarker validation. Neuroimage. 2022 Mar;248:118790. doi: 10.1016/j.neuroimage.2021.118790. Epub 2021 Dec 20. PMID 34933123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was opened in June 2015 and closed in May 2018. First patient enrolled in November 2016 and last enrolled patient completed the study procedures in June 2017. Study enrolled end-of-life subjects (life expectancy less than 6 months) at medical centers in the US who consented to a flortaucipir PET scan and to brain donation at autopsy.
Pre-assignment Details: To be considered eligible for the primary analysis, death had to occur within 6 months of flortaucipir scan and valid autopsy was required.
Groups:
- All Enrolled Cohort: End-of-life subjects (life expectancy < 6 months) consenting to brain donation at autopsy. Subjects will receive a single IV bolus injection of 370 MBq (10 mCi) of flortaucipir.
Period: Overall Study
Arm/Group | All Enrolled Cohort
Started | 3
Completed | 2
Not Completed | 1
Not completed — subject survived greater than 6 months following dosing | 1

BASELINE CHARACTERISTICS:
Population: All subjects consenting to flortaucipir PET and brain donation at autopsy
Groups:
- All Enrolled Cohort: End-of-life subjects (life expectancy < 6 months) consenting to brain donation at autopsy. Subjects received a single IV bolus injection of 370 MBq (10 mCi) of flortaucipir.
Arm/Group | All Enrolled Cohort
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.00 (11.533)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Mini Mental Status Exam (MMSE) Score [Mean (Standard Deviation); unit: units on a scale] — MMSE is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The score ranges from 0 to 30. A score of 23 or lower is indicative of cognitive impairment. Population: n=2 for cognitively impaired subjects. Cognitively normal subject mental status was not measured.
  units on a scale
    number analyzed (Participants) | 2
    (all) | 14.50 (20.5061)
Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) Score [Mean (Standard Deviation); unit: units on a scale] — IQCODE is short questionnaire designed to assess cognitive decline and dementia in elderly people. The questionnaire is filled out by a relative or friend who has known the elderly person for 10 years or more. The result is a score that ranges from 1 to 5. A score of 3 means that the subject is rated on average as 'no change'. A score of 4 means an average of 'a bit worse'. A score of 5 an average of 'much worse'.
  units on a scale | 4.75 (0.4330)

OUTCOME MEASURES:

1. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Whole Cortical Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of whole cortical global quantitation of the PET scan from 82 FreeSurfer-defined regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Groups:
- Autopsy Cohort: End-of-life subjects (life expectancy < 6 months) consenting to brain donation at autopsy. Subjects received a single IV bolus injection of 370 MBq(10 mCi) of flortaucipir and came to autopsy within 6 months of flortaucipir scan.
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | 0.429
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p < 0.001, Spearman's Rank Order Correlation test — A two-sided correlation test (rho ≠ 0) was performed with a significance level of alpha = 0.05 to assess a significant correlation; Correlation coefficient = 0.429

2. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Frontal Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of frontal composite region quantitation of the PET scan regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | 0.681
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p < 0.001, Spearman's Rank Order Correlation test — [p-value comment as in outcome 1, analysis 1]; Correlation coefficient = 0.681

3. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Parietal Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of parietal composite region quantitation of the PET scan regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | 0.644
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p = 0.00278, Spearman's Rank Order Correlation test — [p-value comment as in outcome 1, analysis 1]; Correlation coefficient = 0.644

4. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Cingulate Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of cingulate composite region quantitation of the PET scan regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | 0.437
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p = 0.12, Spearman's Rank Order Correlation test — [p-value comment as in outcome 1, analysis 1]; Correlation coefficient = 0.437

5. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Temporal Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of temporal composite region quantitation of the PET scan regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | 0.324
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p = 0.0712, Spearman's Rank Order Correlation test — [p-value comment as in outcome 1, analysis 1]; Correlation coefficient = 0.324

6. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Occipital Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of occipital composite region quantitation of the PET scan regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | 0.564
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p = 0.0958, Spearman's Rank Order Correlation test — [p-value comment as in outcome 1, analysis 1]; Correlation coefficient = 0.564

7. Primary Outcome: Relationship of Flortaucipir Scan and Pathology - Limbic Composite Region
Description: Correlation between flortaucipir standard uptake value ratio (SUVr) and neuropathology at autopsy. SUVr measurements for the analysis consisted of limbic composite region quantitation of the PET scan regions of interest (ROIs). Values were normalized to the brainstem to obtain the SUVr. Neuropathology was measured by immunohistology using AT8 antibody. Spearman correlation coefficient was calculated. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: autopsy within 6 months of scan
Population: One subject did not come to autopsy within 6 months of the flortaucipir scan.
Measure: Number; unit: Correlation coefficient
Arm/Group | Autopsy Cohort
Number analyzed (Participants) | 2
Correlation coefficient | -0.189
Statistical Analysis 1: Comparison: Autopsy Cohort; Null hypothesis is no correlation (correlation coefficient = 0); Test type: Other; p = 0.558, Spearman's Rank Order Correlation test — [p-value comment as in outcome 1, analysis 1]; Correlation coefficient = -0.189

ADVERSE EVENTS:
Time Frame: Up to a total of 6 months
Description: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. End of study for AE reporting was 48 hours after the last study drug administration. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Groups:
- Safety Analysis Cohort: End-of-life subjects (life expectancy < 6 months) consenting to brain donation at autopsy. Subjects received a single IV bolus injection of 370 MBq (10 mCi) of flortaucipir.
Arm/Group | Safety Analysis Cohort
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The original intent of the protocol was to assess relationships between in vivo flortaucipir PET signal and tau pathology at a higher resolution than the Free Surfer ROIs, such as voxel-wise. Higher resolution could potentially offer more precise insights into tracer distribution patterns. However, the analysis was constrained by challenges in acquiring a complete set of pathology images from collaborators and unanticipated technical challenges in image processing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT02350634/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT02350634/SAP_001.pdf